CLINICAL TRIAL: NCT02295930
Title: Induction Chemotherapy With Folfoxiri Plus Cetuximab and Maintenance With Cetuximab or Bevacizumab Therapy in Unresectable Kras Wild-type Metastatic Colorectal Cancer Patients
Brief Title: Induction Chemoterapy With Folfoxiri Plus Cetuxumab in Unresectable Colorectal Cancer Patient
Acronym: MACBETH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3306; 2011-000840-70 (EudraCT Number)
Record Dates: First submitted 2014-02-04; First posted 2014-11-20 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2015-03

CONDITIONS: Metastatic Colorectal Cancer
Keywords: colorectal cancer,; bevacizumab; cetuximab; folfoxiri; kras wild type
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- folfoxiri+cetuximab+surgery+cetuximab (Experimental): Induction FOLFOXIRI plus cetuximab will consist of:
  * CETUXIMAB 500 mg/sqm IV over 1-h* , day 1 followed by
  * IRINOTECAN 130 mg/sqm IV over 1-h, day 1 followed by
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1 concomitantly with
  * l-LV 200 mg/sqm IV over 2-h, day 1 followed by
  * 5-FLUOROURACIL 2400 mg/sqm IV 48-h continuous infusion, starting on day 1 repeated every 2 weeks for 8 cycles.
  Surgical revaluation will be performed after the induction phase (8 cycles).
  Patients deemed unsuitable for surgery will received maintenance treatment as follows:
  •CETUXIMAB 500 mg/sqm IV over 60-min, day 1 repeated every 2 weeks until PD, patient's refusal, unacceptable toxicity or consent withdrawal.
  Interventions: Other: folfoxiri+cetuximab+surgery+cetuximab
- folfoxiri+cetuximab+surgery+bevacizumab (Experimental): Induction FOLFOXIRI plus cetuximab will consist of:
  * CETUXIMAB 500 mg/sqm IV over 1-h* , day 1 followed by
  * IRINOTECAN 130 mg/sqm IV over 1-h, day 1 followed by
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1 concomitantly with
  * l-LV 200 mg/sqm IV over 2-h, day 1 followed by
  * 5-FLUOROURACIL 2400 mg/sqm IV 48-h continuous infusion, starting on day 1 repeated every 2 weeks for 8 cycles.
  Surgical revaluation will be performed after the induction phase (8 cycles).
  Patients deemed unsuitable for surgery will received maintenance treatment as follows:
  •BEVACIZUMAB 5 mg/kg IV over 30-min, day 1 repeated every 2 weeks until PD, patient's refusal, unacceptable toxicity or consent withdrawal.
  Interventions: Other: folfoxiri+cetuximab+surgery+bevacizumab

INTERVENTIONS:
Other: folfoxiri+cetuximab+surgery+cetuximab — Induction FOLFOXIRI plus cetuximab will consist of:
  * CETUXIMAB 500 mg/sqm IV over 1-h* , day 1 followed by
  * IRINOTECAN 130 mg/sqm IV over 1-h, day 1 followed by
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1 concomitantly with
  * l-LV 200 mg/sqm IV over 2-h, day 1 followed by
  * 5-FLUOROURACIL 2400 mg/sqm IV 48-h continuous infusion, starting on day 1 repeated every 2 weeks for 8 cycles.
  Surgical revaluation will be performed after the induction phase (8 cycles).
  Patients deemed unsuitable for surgery will received maintenance treatment as follows:
  •CETUXIMAB 500 mg/sqm IV over 60-min, day 1 repeated every 2 weeks until PD, patient's refusal, unacceptable toxicity or consent withdrawal.
  Arms: folfoxiri+cetuximab+surgery+cetuximab
Other: folfoxiri+cetuximab+surgery+bevacizumab — Induction FOLFOXIRI plus cetuximab will consist of:
  * CETUXIMAB 500 mg/sqm IV over 1-h* , day 1 followed by
  * IRINOTECAN 130 mg/sqm IV over 1-h, day 1 followed by
  * OXALIPLATIN 85 mg/sqm IV over 2-h, day 1 concomitantly with
  * l-LV 200 mg/sqm IV over 2-h, day 1 followed by
  * 5-FLUOROURACIL 2400 mg/sqm IV 48-h continuous infusion, starting on day 1 repeated every 2 weeks for 8 cycles.
  Surgical revaluation will be performed after the induction phase (8 cycles).
  Patients deemed unsuitable for surgery will received maintenance treatment as follows:
  •BEVACIZUMAB 5 mg/kg IV over 30-min, day 1 repeated every 2 weeks until PD, patient's refusal, unacceptable toxicity or consent withdrawal.
  Arms: folfoxiri+cetuximab+surgery+bevacizumab

SUMMARY:
This is a phase II randomized study of 4-months induction first-line chemotherapy with FOLFOXIRI + cetuximab followed by maintenance with cetuximab or bevacizumab in patients affected by KRAS wild type (wt) mCRC.

DETAILED DESCRIPTION:
The aim of the study is to obtain a rapid disease control with the therapy and the maximum tumoral shrinkage, and than to treat patient with less intensive maintenance to inhibit tumoral regrowth.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma;
* Availability of formalin-fixed paraffin embedded tumor block from primary and/or metastasis;
* KRAS wild-type status of primary colorectal cancer or related metastasis;
* Unresectable and measurable metastatic disease according to RECIST criteria;
* Male or female, aged > 18 years and < 75 years;
* ECOG PS < 2 if aged < 71 years, ECOG PS = 0 if aged 71-75 years;
* Life expectancy of more than 3 months;
* Adequate haematological function: ANC ≥ 1.5 x 109/L; platelets ≥ 100 x 109/L, Hb ≥ 9 g/dL;
* Adequate liver and renal function: serum bilirubin ≤ 1.5 x ULN; alkaline phosphatase and transaminases ≤ 2.5 x ULN (in case of liver metastases < 5 x ULN); serum creatinine ≤ 1.5 x ULN;
* Previous adjuvant chemotherapy containing oxaliplatin is allowed if more than 12 months have elapsed between the end of adjuvant therapy and first relapse;
* Previous adjuvant chemotherapy with fluoropyrimidine monotherapy is allowed if more than 6 months have elapsed between the end of adjuvant and first relapse;
* At least 6 weeks from prior extended radiotherapy and 4 weeks from surgery;
* Written informed consent to experimental treatment and KRAS analysis.

Exclusion Criteria:

* Prior palliative chemotherapy;
* Prior treatment with EGFR or VEGF inhibitors;
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria;
* Presence or history of CNS metastasis;
* Active uncontrolled infections; active disseminated intravascular coagulation;
* Past or current history of malignancies other than colorectal carcinoma, except for curatively treated basal and squamous cell carcinoma of the skin cancer or in situ carcinoma of the cervix;
* Clinically significant cardiovascular disease: cerebrovascular accidents or myocardial infarction ≤ 12 months before treatment start, unstable angina, NYHA ≥ grade 2 chronic heart failure, uncontrolled arrhythmia, uncontrolled hypertension;
* Serious, non-healing wound, ulcer, or bone fracture;
* Evidence of bleeding diathesis or coagulopathy;
* Major surgical procedure or significant traumatic injury within 28 days prior to study treatment start;
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes or chronic, daily treatment with high-dose aspirin (>325 mg/day);
* Subtotal colectomy, malabsorption syndrome and chronic inflammatory bowel disease (i.e. ulcerative colitis, Chron syndrome);
* Fertile women (<2 years after last menstruation) and men of childbearing potential not willing to use effective means of contraception.
* Psychiatric disorder precluding understanding of information on trial related topics,
* Serious underlying medical condition (judged by the investigator) which could impair the ability of the patient to participate in the trial (e.g. uncontrolled diabetes mellitus, active autoimmune disease)
* Concurrent treatment with other experimental drugs or other anti-cancer therapy; treatment in a clinical trial within 30 days prior to trial entry
* Definite contraindications for the use of corticosteroids and antihistamines as premedication
* Known hypersensitivity to trial drugs or hypersensitivity to any other component of the trial drugs
* Any concomitant drugs contraindicated for use with the trial drugs according to the product information of the pharmaceutical companies
* Pregnancy
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial
* Medical or psychological condition which, in the opinion of the investigator, would not permit the patient to complete the study or sign meaningful informed consent

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2011-10; Primary Completion 2015-03 (Actual)

PRIMARY OUTCOMES:
10 months-progression free rate (10m-PFR) | up to 10 months
  10m-PFR is defined as the proportion of patients free from disease progression 10 months after randomization, relative to the total of enrolled patients. Patients whose disease status cannot be evaluated within 11 months after randomization and patients lost to follow up or dead within 10 months after randomization will be considered as progressed for the purpose of the primary endpoint analyses.

SECONDARY OUTCOMES:
Best overall response rate | every 8 weeks, up to 60 months
  Best overall response rate is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements that will be subsequently confirmed by a central review. Responses will be evaluated every 8 weeks until disease progression or up to 60 months. Patients who do not have an on-study assessment will be included in the analysis as non responders.
10 month resection rate | within 10 months after randomization
  10month resection rate is defined as the percentage of patients,relative to the total of enrolled subjects,undergoing secondary R0 resection of metastases within 10months after randomization.Secondary R0 surgery is defined as microscopically margin free complete surgical removal of all residual disease,performed during treatment or after its completion,allowed by tumoral shrinkage and/or disappearance of 1or more lesions.Patients lost to follow up,with disease progression or dead,within 10months after randomization,will be considered as failures.
Time to strategy failure | from randomization, up to 60 months
  It is defined as the time from randomization to one of the followings:
  1. progression during FOLFOXIRI + cetuximab or during a modified FOLFOXIRI + cetuximab regimen;OR
  2. progression and decision to not administer FOLFOXIRI + cetuximab or a modified FOLFOXIRI + cetuximab regimen
  3. introduction of a new agent not included in the study treatment according to randomization arm;OR
  4. death; whichever occurs first.All events will be assessed up to 60 months.For patients still on treatment at the time of analysis, the time to strategy failure will be censored on the last date the patients were known to be alive.
Time to 2nd progressive disease | from randomization, up to 60 months
  It is defined as the time from randomization to 2°documentation of objective disease progression or death due to any cause,whichever occurs first.All events will be assessed up to 60 months.Time to 2nd progressive disease will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive,on study and second progression free at the time of the analysis.Alive patients having no tumor assessments after baseline will have time to event endpoint censored on the date of randomization
Progression free survival (PFS) | from randomization to first documentation of objective disease progression or death, up to 60 months
  It is defined as the time from randomization to first documentation of objective disease progression or death due to any cause,whichever occurs first. All events will be assessed up to 60 months. PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive,on study and progression free at the time of the analysis.Alive patients having no tumor assessments after baseline will have time to event endpoint censored on the date of randomization
Overall survival (OS) | as the time from randomization to the date of death, up to 60 months
  It is defined as the time from randomization to the date of death due to any cause. All events will be assessed up to 60 months. For patients still alive at the time of analysis, the OS time will be censored on the last date the patients were known to be alive.
Toxicity rate | during the induction and the maintenance phases of treatment
  It is defined as the percentage of patients,relative to the total of enrolled subjects,experiencing a specific adverse event of grade 3/4,according to National Cancer Institute Common Toxicity Criteria (version 4.0),during the induction and the maintenance phases of treatment.
Overall toxicity rate | during the induction and the maintenance phases of treatment
  It is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Alfredo Falcone, MD, Principal Investigator — Polo Oncologico Area Vasta Nord Ovest
Locations (22):
- Italy (22):
  - A.O.Universitaria Policlinico S.Orsola-Malpighi Di Bologna (Oncologia Medica), Bologna, Italy
  - AUSL DI FROSINONE - FROSINONE (FR) ONCOLOGIA MEDICA U.O. Oncologia Medica, Frosinone, Italy
  - Ausl 12 Di Viareggio (Lu) - Lido Di Camaiore (Lu) Oncologia Medica, Lucca, Italy
  - AZIENDA OSPEDALIERA DI PERUGIA - OSPEDALE S. MARIA DELLA MISERICORDIA - PERUGIA (PG) ONCOLOGIA MEDICA U.O. Oncologia Medica, Perugia, Italy
  - Polo Oncologico Area Vasta Nord Ovest, Pisa, Italy
  - Ospedale Civile Ss. Antonio E Biagio Di Alessandria - Alessandria (Al) Oncologia Medica, Alessandria
  - Irccs Centro Di Riferimento Oncologico (Cro) - Aviano (Pn), Aviano
  - Istituto Ospedaliero Fondazione Poliambulanza Di Brescia - Brescia (Bs) Oncologia Medica, Brescia
  - Pres.Ospedal.Spedali Civili Brescia - Brescia (Bs) Oncologia Medic, Brescia
  - Ospedale Armando Businco - Cagliari (Ca) Oncologia Medica, Cagliari
  - Azienza Ospedaliera S. Croce E Carle, Cuneo
  - IRCCS ISTITUTO NAZIONALE PER LA RICERCA SUL CANCRO (IST) - GENOVA (GE) ONCOLOGIA MEDICA Oncologia Medica A, Genova
  - Irccs Istituto Oncologico Veneto (Iov) - Padova (Pd) Oncologia Medica, Padua
  - AUSL 5 DI PISA - PISA (PI) ONCOLOGIA MEDICA oncologia medica Osp Lotti Pontedera, Pontedera
  - Ospedale Di S. Maria Nuova - Reggio Nell'Emilia (Re) Oncologia Medica, Reggio Emilia
  - Policlinico Universitario Campus Bio-Medico Di Roma - Roma (Rm) Oncologia Medica, Roma
  - POLICLINICO UMBERTO I DI ROMA - ROMA (RM) ONCOLOGIA MEDICA oncologia Medica, Roma
  - Ospedale Fatebenefratelli, Roma
  - Ospedale San Pietro Fatebenefratelli - Roma (Rm) Oncologia Medica, Roma
  - Ospedale Civile Di Sondrio, Sondrio
  - A.O. Universitaria S. Giovanni Battista-Molinette Di Torino - Torino (to) Oncologia Medica, Torino
  - A.O. UNIVERSITARIA S. MARIA DELLA MISERICORDIA DI UDINE - UDINE (UD) ONCOLOGIA MEDICA U.O. Oncologia Medica, Udine

REFERENCES:
- [Derived] Cremolini C, Antoniotti C, Lonardi S, Aprile G, Bergamo F, Masi G, Grande R, Tonini G, Mescoli C, Cardellino GG, Coltelli L, Salvatore L, Corsi DC, Lupi C, Gemma D, Ronzoni M, Dell'Aquila E, Marmorino F, Di Fabio F, Mancini ML, Marcucci L, Fontanini G, Zagonel V, Boni L, Falcone A. Activity and Safety of Cetuximab Plus Modified FOLFOXIRI Followed by Maintenance With Cetuximab or Bevacizumab for RAS and BRAF Wild-type Metastatic Colorectal Cancer: A Randomized Phase 2 Clinical Trial. JAMA Oncol. 2018 Apr 1;4(4):529-536. doi: 10.1001/jamaoncol.2017.5314. PMID 29450468